CLINICAL TRIAL: NCT00536705
Title: Effect of Montelukast on the Expression and Variation of TGF-β for Children With Mild Persistent Asthma
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: The first people's hospital of shanghai, department of pediatric
Other Study IDs: #p2192v1
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2009-01

CONDITIONS: Asthma
Keywords: asthma; child; transforming growth factor beta(TGF-β); Leukotriene Antagonists(Montelukast)
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subjects inhaled hypertonic saline (3%) via an ultrasonic nebulizer with the output set at maximum for 20 minutes. To collect sputum, subjects were asked to expectorate the sputum onto a plastic Petri dish after the 20-min period of inhalation. During the inducing procedure, macroscopic characteristics of the sputum were recorded and adequate plugs of sputum were separated from saliva and processed immediately after expectoration.The complete blood count, platelet count, and serum biochemical analyses were done meanwhile.

INTERVENTIONS:
Drug: montelukast — montelukast 5-mg chewable tablet with matching placebo once daily in the evening at bedtime.The study consisted of a 2-week, single-blind placebo baseline period and a 12-week double-blind, active treatment period
  Other Names: singulair

SUMMARY:
The Objective of our research is to observe the effect of cysteinyl leukotriene receptor antagonist on the expression and variation of TGF-β1 levels and mRNA expression in children with mild persistent asthma in their plasma and T lymphocyte, to discuss the role of TGF-β1 in the pathogenesis of bronchial asthma in children and to evaluate the function of regulation of leukotriene receptor antagonist on asthma in children.

DETAILED DESCRIPTION:
The majority pediatric asthma patients in Shanghai are mild persistent asthma. These patients require controller medications every day to achieve and maintain control. Leukotriene receptor antagonist is one of the options which have been recommended to use as a mono controller therapy. Patient satisfaction and compliance was better with montelukast, attributed to oral intake and convenience. Owing to its easy and simple oral once a day administration montelukast was found to be advantageous over ICS. On the other hand, recent studies have shown that there is a considerable degree of airway remodeling in peripheral airways in patients with mild asthma.The new information points out the need for large, long term studies on the treatment of mild persistent asthma, with an emphasis on exacerbations, remodeling, and the relationship between these outcomes and markers of asthma control. TGF-β participates in the initiation and propagation of inflammatory and immune responses in the airways. The leukotrienes exert their biologic actions by binding to and activating specific receptors. Montelukast, a cysteinyl leukotriene 1(CysLT1) receptor antagonist, acts on LTC4, LTD4 and LTE4, and, therefore, on airway inflammation and bronchoconstriction. Some results suggest that low dose of Montelukast may modulate the parameters of inflammation and fibrosis.In this study we try to determine the effects of lower dose Montelukast on the expression and variation of TGF-β in induced sputum and T lymphocyte for children with mild persistent Asthma.

Drug in the study provide by MSD. We have done induced sputum procedure in our past study. Reagent can be bought from company.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 to 14 years with a history of physician-diagnosed asthma (at least 3 episodes of asthma symptoms during the previous year, including, but not limited to cough, wheezing, and shortness of breath)

Exclusion Criteria:

* Patients were not in good health, other than asthma, on the basis of results of medical history, physical examination, and routine laboratory tests.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: After screening 200 patients, we randomized 120 patients aged 6 to 14 years with a history of physician-diagnosed asthma .These patients randomized into montelukast group and placebo group.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: hong jianguo, prof, Principal Investigator — pediatric of shanghai jiantong University
Locations (1):
- Shanghai First People'S Hospital, Shanghai, Shanghai Municipality, China